CLINICAL TRIAL: NCT03592251
Title: Efficacy Evaluation of 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Memory Consolidation in Healthy Adults
Brief Title: 26 Weeks' Dietary Supplementation With DHA- and EPA-enriched Oils on Memory Consolidation in Healthy Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northumbria University (Other)
Collaborators: BASF (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 44N6
Record Dates: First submitted 2018-05-29; First posted 2018-07-19 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Memory Consolidation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Olive oil Placebo (Placebo Comparator): 3 x 1 g capsules daily Placebo: olive oil
  Interventions: Dietary Supplement: EPA-rich; Dietary Supplement: DHA-rich
- EPA-rich (Active Comparator): 3 x 1 g capsules daily containing a SMEDDS formulation of an EPA-enriched oil totalling 900 mg EPA and 360 mg of DHA
  Interventions: Dietary Supplement: Olive Oil Placebo; Dietary Supplement: DHA-rich
- DHA-Rich (Active Comparator): 3 x 1 g capsules daily containing a SMEDDS formulation of an DHA-enriched oil totalling 900 mg DHA and 270 mg of EPA
  Interventions: Dietary Supplement: Olive Oil Placebo; Dietary Supplement: EPA-rich

INTERVENTIONS:
Dietary Supplement: Olive Oil Placebo — 6 months placebo supplementation
  Arms: DHA-Rich; EPA-rich
Dietary Supplement: EPA-rich — 6 months placebo supplementation
  Arms: DHA-Rich; Olive oil Placebo
Dietary Supplement: DHA-rich — 6 months placebo supplementation
  Arms: EPA-rich; Olive oil Placebo

SUMMARY:
The purpose of this study is to investigate the effects of EPA- and DHA-enriched omega-3 polyunsaturated fatty acid dietary supplements on overnight verbal and visual memory consolidation as well as morning alertness before and after 26 weeks of supplementation

ELIGIBILITY:
Inclusion Criteria:

* Aged 25 to 49 years inclusive
* Males and females
* Self-report of good health

Exclusion Criteria:

* English is not first language (some of the cognitive tasks have only been validated in native English speakers)
* Habitual consumption of oily fish exceeds one fish meal per week
* Habitual consumption of n-3 dietary supplements in the previous 6 months
* Habitual use of dietary supplements within the last month (defined as more than 3 consecutive days or 4 days in total; some supplements that do not impact upon cognitive function e.g. garlic, protein, calcium are allowed. Please check with the research team if you are unsure)
* Are a smoker or consume any nicotine replacement products (e.g. chewing gum, e-cigarettes)?
* Food allergies or sensitivities to any of the ingredients contained in the investigational product or any other foodstuff
* Pregnant, trying to get pregnant or breast feeding
* Body Mass Index outside of the range 18-35 kg/m2
* High blood pressure (systolic over 159 mm Hg or diastolic over 99 mm Hg)
* Currently taking blood pressure medication
* Currently taking blood thinning medication (e.g. aspirin, warfarin, heparin)
* Have a respiratory disorder that requires regular medication (Note: participants with asthma who only take their medication occasionally/as required are eligible for this study)
* Have frequent migraines that require medication (more than or equal to 1 per month)
* History or current diagnosis of drug/alcohol abuse
* History of kidney or liver disease, or other severe diseases of the gastrointestinal tract (e.g. iron accumulation, iron utilization disorders, hypercalcaemia, hypercalcaemia), that are likely to interfere with metabolism/absorption/secretion of the product under investigation
* History of neurological or psychiatric illness (excluding depressive illness and anxiety)
* History of head trauma
* Sleep disturbances and/or are taking sleep aid medication
* Blood disorders (e.g. anaemia, haemophilia, thrombocytosis)
* Diagnosis of type I or type II diabetes
* Heart disorder, or vascular illness
* Current diagnosis of depression and/or anxiety
* Over- or under-active thyroid
* Chronic gastrointestinal problems (e.g. Inflammatory Bowel Disease, Irritable Bowel Syndrome, celiac disease)
* Any known active infections
* Diagnosed with or may be at risk of having syphilis, hepatitis, the Human T - lymphotropic virus or the Human Immunodeficiency Virus
* Current or past breast cancer diagnosis and/or a mastectomy
* Health condition that would prevent fulfilment of the study requirements
* Currently participating in or in the past 4 weeks participated in other clinical or nutrition intervention studies

Ages: 25 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Computerised Location Learning task | 26 months
  Delayed recall accuracy
Verbal Learning task | 26 months
  Delayed recall accuracy

SECONDARY OUTCOMES:
Computerised Location Learning task | 26 months
  Learning index
Verbal Learning task | 26 months
  Learning index
Peg and Ball/Tower of London task | pre, Mid and post dose measures
  Planning time (ms)
Peg and Ball/Tower of London task | pre, Mid and post dose measures
  Completion time (ms)
Peg and Ball/Tower of London task | pre, Mid and post dose measures
  Errors (number)
Simple reaction time task | 26 months
  reaction time speed from a simple reaction task
Digit vigilance task | 26 months
  accuracy (%)
Digit vigilance task | 26 months
  Reaction time (ms)
Subjective Alertness | 26 months
  Subjective ratings of alertness upon waking on a visual analogue scale (0-100 with 100 denoting the most alert the participant has ever felt in their life)

CONTACTS AND LOCATIONS:
Locations (1):
- Northumbria University, Newcastle upon Tyne, Tyne and Wear, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patan MJ, Kennedy DO, Husberg C, Hustvedt SO, Calder PC, Khan J, Forster J, Jackson PA. Supplementation with oil rich in eicosapentaenoic acid, but not in docosahexaenoic acid, improves global cognitive function in healthy, young adults: results from randomized controlled trials. Am J Clin Nutr. 2021 Sep 1;114(3):914-924. doi: 10.1093/ajcn/nqab174. PMID 34113957